CLINICAL TRIAL: NCT03683498
Title: A Phase I Trial of Donor Regulatory T-cells for Steroid-Refractory Chronic Graft-versus-Host-Disease in Patients Who do Not Obtain Complete Remission With Ruxolitinib
Brief Title: Donor Regulatory T-cells for Steroid-Refractory Chronic Graft-versus-host-Disease
Acronym: GVHD-TReG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GVHD-TReG
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Chronic Graft vs Host Disease
Keywords: Ruxolitinib; T cells

STUDY DESIGN:
Intervention Model Description: Initial enrollment will be at Dose-level A. Subsequent cohorts will be dose escalated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regulatory T-cell enriched infusion (Experimental): Dose escalation sequential cohorts Regulatory T-cell enriched infusion (Cells/kg) will be administered. The cohorts will be dose escalated per the schema below:
  Dose-level A: 0.5 x 10ˆ6 Cells/kg Dose-level B: 1 x 10ˆ6 cell/kg Dose-level C: 2 x 10ˆ6 cell/kg
  Interventions: Biological: Regulatory T-cell enriched infusion

INTERVENTIONS:
Biological: Regulatory T-cell enriched infusion — Enrichment of CD25hi regulatory T cells from CD8 and/or CD19 pre-depleted leukapheresis products.

SUMMARY:
A Phase I Trial of Donor Regulatory T-cells for Steroid-Refractory Chronic Graft-versus-Host-Disease in patients who do not obtain complete remission with ruxolitinib

DETAILED DESCRIPTION:
The study design is based on a phase I trial in Spanish.

A number of 16 patients will be included to assess the safety and maximum tolerated dose-level of donor regulatory enriched T cell (Treg) in steroid-refractory chronic graft versus host disease (cGVHD) patients who did not obtain complete remission under treatment with ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of allogeneic hematopoietic stem cell transplantation.
* Participants must have steroid-refractory cGVHD and had obtained a partial response after at least 4 weeks of treatment with ruxolitinib.
* Steroid-refractory cGVHD is defined as having persistent signs and symptoms of cGVHD (Appendix D) despite the use of prednisone at ≥0.25 mg/kg/day (or 0.5 mg/kg every other day) for at least 4 weeks (or equivalent dosing of alternate glucocorticoids) without complete resolution of signs and symptoms.
* Stable dose of glucocorticoids for 4 weeks prior to enrolment
* No addition or subtraction of other immunosuppressive medications (e.g., calcineurin-inhibitors, sirolimus, mycophenolate-mofetil) for 4weeks prior to enrolment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug
* No age limit. In the case of children participating in the study, the informed consent will be signed by a parents or legal guardians
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Participants must have adequate organ function
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Ongoing prednisone requirement >1 mg/kg/day (or equivalent).
* Concurrent use of calcineurin-inhibitor plus sirolimus (either agent alone is acceptable).
* History of thrombotic microangiopathy, hemolytic-uremic syndrome or thrombotic thrombocytopenic purpura.
* New immunosuppressive medication in the 4 weeks prior.
* Extra-corporeal Photopheresis or rituximab therapy in the 4 weeks prior.
* Post-transplant exposure to T-cell or Interleukin-2 targeted medication (e.g. alemtuzumab, basiliximab, denileukin diftitox) within 100 days prior.
* Donor lymphocyte infusion within 100 days prior.
* Active malignant relapse.
* Active uncontrolled infection.
* Organ transplant (allograft) recipient.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the agents used after allogeneic hematopoietic stem cell transplant (HSCT). In addition, these individuals are at increased risk of lethal infections. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Individuals with active uncontrolled hepatitis B or C are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after hematopoietic stem cell transplant (HSCT).
* Other investigational drugs within 4 weeks prior to enrolment, unless cleared by the Principal Investigator.
* Pregnant women are excluded from this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Toxicity and maximum tolerated dose | Up 12 weeks after infusion
  To determine the maximum tolerated dose (MTD) and toxicity of Treg-enriched infusion among patients receiving ruxolitinib.

SECONDARY OUTCOMES:
Quantification of targeted cells of manufacturing Treg-enriched product meeting the targeted cell dose-level. | Before 24 hours to infusion up infusion day
  Percentage of cells viability, negative gram stain/endotoxin, percentage of CD4+CD25+ cells and CD4+CD25+CD127- Treg in order to consider for the infusion.
Clinical response of Treg-enriched infusion | Up 12 weeks after Treg infusion
  Each participant should be assigned one of the following categories: 1) complete cGVHD response per NIH criteria, 2) partial cGVHD response per NIH criteria, 3) non-response (includes stable disease) per NIH criteria, 4) progressive cGVHD per NIH criteria, 5) malignant disease relapse, or 6) unknown (not assessable, insufficient data).
Immunologic effects through phenotypical evaluation | Up 12 weeks after Treg infusion
  Phenotypical evaluation of T cell populations (CD4, CD8, Treg), B and NK cells nuclear cells of Treg-enriched infusion among patients receiving ruxolitinib.
Immunologic effects through immune globulins. | Up 12 weeks after Treg infusion
  Quantitative immune globulins of Treg-enriched infusion among patients receiving ruxolitinib
Immunologic effects through plasma banking | Up 12 weeks after Treg infusion
  Plasma banking of Treg-enriched infusion among patients receiving ruxolitinib
Immunologic effects through additional mononuclear cells. | Up 12 weeks after Treg infusion
  Storage of additional mononuclear cells of Treg-enriched infusion among patients receiving ruxolitinib
Survival after one year of Treg infusion | 1 year after Treg infusion
  Number of patients alive after one year of Treg infusion

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pérez-Simón, M.D. Ph.D., Principal Investigator — Department of Hematology, Hospital Universitario Virgen del Rocío, Sevilla.
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soares MV, Escamilla Gomez V, Azevedo RI, Pereira PNG, Caballero-Velazquez T, Mendes L, Alho AC, Garcia-Guerrero E, Garcia-Calderon CB, Tharmaratnam K, Cabral IA, Ribeiro AC, Juncal C, Roncon S, Pais AT, Rodriguez-Gil A, Espada ELDS, Rodrigues A, Garcao A, Yaspo ML, Warnatz HJ, Lehrach HR, Ward L, Barbosa-Morais NL, Quintas AM, Palmela P Sr, Caldas CMF, Ferreira R, Leite L, Martins C, Lourenco F, Moreno R, Campilho F, Cheyne CP, Garcia-Finana M, Campos AM, Baron F, Arpinati M, Hoffmann P, Edinger M, Koreth J, Ritz J, Pinho Vaz C, Perez-Simon JAA, Lacerda JF. Phase I/II Trials of Donor Regulatory T Cells for the Treatment of Steroid-Refractory Chronic Graft versus Host Disease. Blood Adv. 2026 Feb 4:bloodadvances.2025017996. doi: 10.1182/bloodadvances.2025017996. Online ahead of print. PMID 41637631